CLINICAL TRIAL: NCT02067611
Title: A Phase 2, Multicenter, Randomized, Double Blind, Placebo Controlled, Parallel Group, Dose Range Finding Study to Evaluate the Efficacy and Safety of X0002 Spray Versus Placebo in Subjects With Osteoarthritis
Brief Title: A Study to Evaluate the Efficacy and Safety of X0002 Spray in Subjects With Osteoarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lina Xu (Industry)
Responsible Party: Sponsor-Investigator, Lina Xu, Vice president, Techfields Pharma Co. Ltd
Organization: Techfields Pharma Co. Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TF-X0002-21
Record Dates: First submitted 2014-02-18; First posted 2014-02-20 (Estimated); Results first posted 2018-02-07 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Osteoarthritis of the Knee
Keywords: Phase 2, Efficacy, Safety, Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Bulk Drugs

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- X0002 (Experimental): low dose, BID;middle dose, BID, or high dose, BID.
  Interventions: Drug: X0002
- Placebo (Placebo Comparator): low dose, BID; middle dose, BID, or high dose, BID.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: X0002 — Parallel Assignment
  Other Names: Active drug
  Arms: X0002
Drug: Placebo — Parallel Assignment
  Other Names: Placebo powder
  Arms: Placebo

SUMMARY:
This is a phase 2, multicenter, randomized, double blind (with dose), placebo controlled, parallel group, proof of concept, and dose range finding study to evaluate the efficacy, safety, and PK of X0002 spray in adult subjects with clinically symptomatic mild to moderate OA of the knee.

Objectives of the study:

1. To evaluate the efficacy of X0002 spray compared to placebo for relief of knee pain in subjects with osteoarthritis (OA) of the knee;
2. To assess the safety and tolerability of multiple doses of X0002 when administered as a topical spray.

DETAILED DESCRIPTION:
This is a phase 2, multicenter, randomized, double blind (with dose), placebo controlled, parallel group, proof of concept, and dose range finding study to evaluate the efficacy, safety, and PK of X0002 spray in adult subjects with clinically symptomatic mild to moderate OA of the knee.

After a screening period of up to 3 weeks and radiographic evaluation of the target knee joint space, 225 subjects will be randomly assigned to 1 of 3 treatment groups in a 1:1:1 ratio with a 2:1 ratio of active:placebo within each treatment group in a 1:1:1 ratio with a 2:1 ratio of active:placebo within each treatment group (i.e., 2 subjects to active treatment and 1 subject to placebo):

Group A: low dose of X0002, twice daily (BID, approximately every 12 hours; n=50) or placebo (low dose), BID (approximately every 12 hours; n=25); Group B: middle dose of X0002, BID (approximately every 12 hours; n=50) or placebo , BID (approximately every 12 hours; n=25) ; Group C: High dose of X0002, BID (approximately every 12 hours; n=50) or placebo, BID (approximately every 12 hours; n=25) .

Safety and efficacy assessments will be performed at at 2, 4, 8, and 12 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* A subject must be a male or female between 35 and 85 years of age, inclusive.
* A subject must have a body mass index (BMI) between 18.5 and 39.9 kg/m2, inclusive.
* A subject must have a diagnosis of idiopathic OA according to the American College of Rheumatology (ACR) clinical and radiographic criteria (knee pain, osteophytes, and at least one of the following: >50 years of age, morning stiffness lasting <30 minutes after getting up in the morning, or crepitus).
* A subject must have a Kellgren Lawrence Grade of 1 or 2 as determined by the Investigator or a local radiologist at Screening.
* A subject must have a history of clinically symptomatic mild to moderate OA of the knee for ≥6 months.
* A subject must have had knee pain while standing, walking, and/or on motion for at least 14 days during the month prior to Screening.
* A subject must have a knee pain score ≥40 mm and <90 mm on a 100 mm VAS (with or without analgesic medication) on at least 10 of the 14 days prior to randomization.
* A subject must be willing to discontinue any NSAIDs or other analgesic (eg, aspirin, acetaminophen) or potentially confounding concomitant treatments (eg, physiotherapy, acupuncture) starting 4 days before the administration of the first dose of study medication until completing participation in the study. (The use of ≤325 mg acetylsalicylic acid per day as cardiac prophylaxis is permitted.) The subject will be allowed to take rescue medication (acetaminophen) for pain during the study except during the 24 hours prior to Baseline (Day1), Week 2, Week 4, Week 8, Week 12/EOS, and Follow-up assessments.
* A subject must be willing to avoid unaccustomed physical activity (eg, starting a new weight lifting routine) for the duration of the study.

Exclusion Criteria:

* A subject who has secondary OA of the knee or OA of lower limb joints other than the knee that, in the opinion of the Investigator, could interfere with pain and functional assessments related to the knee
* A subject who has OA of the knee with a Kellgren Lawrence Grade ≥3 as determined by the Investigator or a local radiologist at Screening
* A subject who has a history of total or partial knee replacement, arthroplasty, or other knee surgery on either knee
* A subject who has had significant injury, as judged by the Investigator, involving the target knee within the 6 months before Screening.
* A subject who has skin lesions or wounds on or near the knees to be treated at Screening or on Day 1 prior to the first administration of study medication
* A subject who has used opiates or corticosteroids within 30 days before Screening or who requires treatment with chronic opiates or corticosteroids
* A subject who has had intra articular injections of corticosteroids, hyaluronic acid, or viscosupplements (eg, Synvisc®) to a knee to be treated within the 3 months before Screening.
* A subject who has a history of significant hypersensitivity, intolerance, or allergy to ibuprofen, any NSAIDs, aspirin, or acetaminophen
* A subject who has had an active peptic ulceration in the 12 months prior to Screening or a history of gastrointestinal (GI) bleeding within 5 years of Screening
* A subject who has used an anticoagulant (except aspirin up to 325 mg/day for cardiac prophylaxis) in the month prior to Screening
* A subject who has positive results on fecal occult blood testing at Screening or on Day 1 prior to the first administration of study medication
* A subject who has a history of chronic inflammatory disease (such as rheumatoid arthritis, psoriatic arthritis, gouty arthritis), fibromyalgia, conditions that may affect the target joint (eg, osteonecrosis, chondrocalcinosis), or asthma.

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2014-02; Primary Completion 2015-08 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chongxi Yu, Ph.D., Study Chair — Techfields Inc
Locations (20):
- United States (20):
  - Fiel Family & Sports Medicine/Clinical Research Advantage Inc, Tempe, Arizona
  - Med Center, Carmichael, California
  - Encompass Clinical Research, Spring Valley, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - New England Research Assoc., Trumbull, Connecticut
  - Clinical Research of South Florida, Coral Gables, Florida
  - Avail Clinical Research, LLC, DeLand, Florida
  - Health Awareness Inc., Jupiter, Florida
  - Suncoast Clinical Research, Inc, New Port Richey, Florida
  - Columbus Regional Research Institute, Columbus, Georgia
  - Clinical Trials Technology(CTT) Consultants, Inc., Prairie Village, Kansas
  - Healthcare Research Network, Hazelwood, Missouri
  - Sundance Clinical Research, LLC, St Louis, Missouri
  - New Mexico Clinical Research & Osteoporosis Center, Inc., Albuquerque, New Mexico
  - Hightop Medical Research, Cincinnati, Ohio
  - Prestige Clinical Research, LLC, Franklin, Ohio
  - Heritage Valley Medical Group, Beaver, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Quality Research Inc, San Antonio, Texas
  - Health Research of Hampton Roads, Inc, Newport News, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: Low dose of X0002/placebo, twice per day
- Group B: Middle dose of X0002/placebo, twice per day.
- Group C: High dose of X0002/placebo, twice per day.
Period: Overall Study
Arm/Group | Group A | Group B | Group C
Started | 72 | 72 | 72
Completed | 66 | 66 | 68
Not Completed | 6 | 6 | 4

BASELINE CHARACTERISTICS:
Population: In the study, the active drug and placebo were mixed up and we did not have safety and efficacy data and no report at all.
Groups:
- X0002+Placebo: low dose, BID;middle dose, BID, or high dose, BID.
Arm/Group | X0002+Placebo
Number analyzed (Participants) | 216
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: In this study, the active drug and placebo were mixed up and we did not have safety and efficacy data and no report at all.
Sex: Female, Male [Count of Participants; unit: Participants] — Population: In this study, the active drug and placebo were mixed up and we did not have safety and efficacy data and no report at all.

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate the Efficacy of X0002 Spray Compared to Placebo for Relief of Knee Pain in Subjects With Osteoarthritis (OA) of the Knee
Description: The Primary Efficacy Endpoint is change from Baseline in the WOMAC (VAS) pain subscale score for the target knee at 4 weeks of treatment, and will be analyzed using an analysis of covariance (ANCOVA). Treatment will be included as a fixed class effect and WOMAC Baseline pain subscale score as covariates. The primary comparisons of interest will be the difference between active Group A (low dose) and combined placebo, active Group B (middle dose) and combined placebo, and active Group C (high dose) and combined placebo.
  Safety analyses will be conducted on the SAS. Safety parameters will be listed and summarized using standard descriptive statistics, as appropriate. No formal statistical analyses are planned.
Time Frame: 4 weeks of treatment
Population: The labels for X0002 and placebo were mixed up, and the data was mixed up totally.
Groups:
- Placebo: Low dose, BID; Middle dose, BID; High dose BID
Arm/Group | X0002 | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: To Assess the Safety and Tolerability of Multiple Doses of X0002 When Administered as a Topical Spray
Description: A sensitivity analysis will also be conducted on the Primary Efficacy Endpoint using an ANCOVA with treatment as a fixed class effect and WOMAC baseline pain subscale score as covariates, but the comparisons of interest will be the difference between the active and placebo subjects within each treatment group.
  The Secondary Efficacy Endpoints, change from Baseline in the WOMAC subscale scores for pain, stiffness, and functional ability, and overall WOMAC score at 2, 8, and 12 weeks of treatment, will be by analyzed using the same methods as the for the Primary Efficacy Endpoint.
  Safety analyses will be conducted on the SAS. Safety parameters will be listed and summarized using standard descriptive statistics, as appropriate. No formal statistical analyses are planned.
Time Frame: 2, 8, and 12 weeks of treatment
Population: The labels for X0002 and placebo were mixed up, and the data was mixed up totally.
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: To Evaluate the Effect of X0002 Spray Compared to Placebo for the Relief of Joint Stiffness
Description: A sensitivity analysis will also be conducted on the Primary Efficacy Endpoint using an ANCOVA with treatment as a fixed class effect and WOMAC baseline pain subscale score as covariates, but the comparisons of interest will be the difference between the active and placebo subjects within each treatment group.
  The Secondary Efficacy Endpoints, change from Baseline in the WOMAC subscale scores for pain, stiffness, and functional ability, and overall WOMAC score at 2, 4, 8, and 12 weeks of treatment, will be by analyzed using the same methods as the for the Primary Efficacy Endpoint.
  Safety analyses will be conducted on the SAS. Safety parameters will be listed and summarized using standard descriptive statistics, as appropriate. No formal statistical analyses are planned.
Time Frame: 2, 4, 8, and 12 weeks of treatment
Population: The labels for X0002 and placebo were mixed up, and the data was mixed up totally.
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: To Assess the Effect of X0002 Spray Compared to Placebo on Difficulty Performing Daily Activities
Description: as for outcome 2
Time Frame: at 2, 4, 8, and 12 weeks of treatment
Population: The labels for X0002 and placebo were mixed up, and the data was mixed up totally.
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Characterize the Pharmacokinetics of X0002
Description: Cmax, Tmax, AUCs, apparent terminal elimination rate constant, apparent terminal elimination half-life will be calculated.
Time Frame: at the Week 2, week 3, week 4 and Week 12
Population: The labels for X0002 and placebo were mixed up, and the data was mixed up totally.
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 0 | 0 | 0

6. Other Pre Specified Outcome: Subject's Global Assessment of Disease Status of the Target Knee at 2, 4, 8 and 12 Weeks of Treatment
Description: Data for the exploratory efficacy endpoints will be summarized using descriptive statistics.
  Safety analyses will be conducted on the SAS. Safety parameters will be listed and summarized using standard descriptive statistics, as appropriate. No formal statistical analyses are planned.
Time Frame: at 2, 4, 8, and 12 weeks of treatment
Population: The labels for X0002 and placebo were mixed up, and the data was mixed up totally.
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 0 | 0 | 0

7. Other Pre Specified Outcome: Investigator's Global Assessment of Disease Status of the Target Knee at 2, 4, 8 and 12 Weeks of Treatment
Description: as for outcome 6
Time Frame: at 2, 4, 8, and 12 weeks of treatment
Population: The labels for X0002 and placebo were mixed up, and the data was mixed up totally.
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 0 | 0 | 0

8. Other Pre Specified Outcome: Subject's Global Assessment of Response to Therapy of the Target Knee at 2, 4, 8 and 12 Weeks of Treatment
Description: as for outcome 6
Time Frame: at 2, 4, 8, and 12 weeks of treatment
Population: The labels for X0002 and placebo were mixed up, and the data was mixed up totally.
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 0 | 0 | 0

9. Other Pre Specified Outcome: Investigator's Global Assessment of Response to Therapy of the Target Knee at 2, 4, 8 and 12 Weeks of Treatment
Description: as for outcome 6
Time Frame: at 2, 4, 8, and 12 weeks of treatment
Population: The labels for X0002 and placebo were mixed up, and the data was mixed up totally.
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 0 | 0 | 0

10. Other Pre Specified Outcome: Change From Baseline Over Time in VAS Pain Scores for the Target Knee From Daily Diary Data.
Description: as for outcome 6
Time Frame: at 2, 4, 8, and 12 weeks of treatment
Population: The labels for X0002 and placebo were mixed up, and the data was mixed up totally.
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 0 | 0 | 0

11. Other Pre Specified Outcome: Amount of Rescue Medication (Acetaminophen) Consumed Per Day for Target Knee Pain.
Description: as for outcome 6
Time Frame: at 2, 4, 8, and 12 weeks of treatment
Population: The labels for X0002 and placebo were mixed up, and the data was mixed up totally.
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: This study was ongoing for about 16 weeks (12 weeks treatment, 1 week follow-up and 3 weeks screening). Safety assessments were performed at each visit and included assessment of AEs, vital signs (blood pressure, pulse rate, and oral temperature), clinical laboratories, physical examination, skin irritation, and electrocardiograms (ECGs).
Description: In this study, the active drug and placebo were mixed up and we did not have safety and efficacy data and no report at all.
Groups:
- X0002/Placebo: low dose, BID;middle dose, BID, or high dose, BID.
Arm/Group | X0002/Placebo
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes